CLINICAL TRIAL: NCT00384176
Title: A Randomised, Double-blind, Multicentre Phase II/III Study to Compare the Efficacy of Cediranib (RECENTIN™, AZD2171) in Combination With 5-fluorouracil, Leucovorin, and Oxaliplatin (FOLFOX), to the Efficacy of Bevacizumab in Combination With FOLFOX in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: First Line Metastatic Colorectal Cancer Therapy in Combination With FOLFOX
Acronym: HORIZON III
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00013; Eudract Number 2005-003440-66
Record Dates: First submitted 2006-10-03; First posted 2006-10-05 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; RECENTIN
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cediranib; Bevacizumab; Fluorouracil; Folfox protocol; Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Bevacizumab + FOLFOX
  Interventions: Drug: Bevacizumab; Drug: 5-fluorouracil ( in FOLFOX); Drug: Leucovorin (in FOLFOX); Drug: Oxaliplatin (in FOLFOX)
- 2 (Experimental): Cediranib + FOLFOX
  Interventions: Drug: Cediranib; Drug: 5-fluorouracil ( in FOLFOX); Drug: Leucovorin (in FOLFOX); Drug: Oxaliplatin (in FOLFOX)

INTERVENTIONS:
Drug: Cediranib — oral tablet once daily
  Other Names: RECENTIN™; AZD2171
  Arms: 2
Drug: Bevacizumab — intravenous infusion
  Other Names: Avastin®
  Arms: 1
Drug: 5-fluorouracil ( in FOLFOX) — intravenous infusion
  Other Names: 5-FU
Drug: Leucovorin (in FOLFOX) — intravenous infusion
Drug: Oxaliplatin (in FOLFOX) — intravenous infusion
  Other Names: Eloxatin®

SUMMARY:
The purpose of this study is to see if Cediranib in combination with FOLFOX is effective in treating metastatic colorectal cancer and to see how it compares with Avastin (Bevacizumab) in combination with FOLFOX.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of colon or rectal cancer
* No prior systemic therapy for metastatic disease. Any adjuvant/neoadjuvant oxaliplatin therapy must have been received >12 months prior to study entry and adjuvant/neoadjuvant 5-FU must have been received >6 months prior to study entry.

Exclusion Criteria:

* Prior treatment with a VEGF Inhibitor, including bevacizumab and cediranib.
* Poorly controlled hypertension

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1814 (Actual)
Dates: Start 2006-08-30 (Actual); Primary Completion 2009-11-15 (Actual); Study Completion 2015-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca
Locations (280):
- United States (44):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Casa Grande, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Palm Springs, California
  - Research Site, San Diego, California
  - Research Site, Fairfield, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Bay Pines, Florida
  - Research Site, Fort Meyers, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Galesburg, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Layfayette, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, Alexandria, Louisiana
  - Research Site, Layfayette, Louisiana
  - Research Site, Hagerstown, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Summit, New Jersey
  - Research Site, Fresh Meadows, New York
  - Research Site, Northport, New York
  - Research Site, Rochester, New York
  - Research Site, Fayetteville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Coos Bay, Oregon
  - Research Site, Hilton Head Island, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, White River Junction, Vermont
  - Research Site, Abingdon, Virginia
  - Research Site, Alexandria, Virginia
- Australia (40):
  - Research Site, Armidale, New South Wales
  - Research Site, Coffs Harbour, New South Wales
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Hornsby, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Port Macquarie, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Tamworth, New South Wales
  - Research Site, Waratah, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Bedford Park, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Hobart, Tasmania
  - Research Site, Epping, Victoria
  - Research Site, Ashford
  - Research Site, Bedford Park
  - Research Site, Bendigo
  - Research Site, Box Hill
  - Research Site, Camperdown
  - Research Site, Coffs Harbour
  - Research Site, Darlinghurst
  - Research Site, East Melbourne
  - Research Site, Epping
  - Research Site, Herston
  - Research Site, Hobart
  - Research Site, Hornsby
  - Research Site, Kogarah
  - Research Site, Lismore
  - Research Site, Malvern
  - Research Site, Nedlands
  - Research Site, Port Macquarie
  - Research Site, Randwick
  - Research Site, South Brisbane
  - Research Site, St Leonards
  - Research Site, Tamworth
  - Research Site, Waratah
  - Research Site, Wodonga
  - Research Site, Woodville South
- Austria (7):
  - Research Site, Kundratstrasse 3, Vienna
  - Research Site, Innsbruck
  - Research Site, Kundratstrasse 3
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
  - Research Site, Zams
- Belgium (15):
  - Research Site, Bonheiden, Belgium
  - Research Site, Brussels (woluwe-st-lambert), Belgium
  - Research Site, Edegem, Belgium
  - Research Site, Ghent, Belgium
  - Research Site, Kortrijk, Belgium
  - Research Site, Leuven, Belgium
  - Research Site, Roeselare, Belgium
  - Research Site, Bonheiden
  - Research Site, Bruges
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Roeselare
- Canada (16):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, York, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Montreal
- Czechia (6):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Kutná Hora
  - Research Site, Nová Ves pod Pleší
  - Research Site, Pardubice
  - Research Site, Tábor
- Egypt (2):
  - Research Site, Alexandria
  - Research Site, Cairo
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vaasa
- France (6):
  - Research Site, Boulogne
  - Research Site, La Roche S YON
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Saint-Grégoire
- Germany (9):
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, München
  - Research Site, Neu-Isenburg
  - Research Site, Tübingen
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Tatabánya
- India (14):
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Varanasi, Uttar Prad
  - Research Site, Kolkata, West Bengal
  - Research Site, Bangalore
  - Research Site, Bhopal
  - Research Site, Chennai
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Pune
  - Research Site, Sheikhpura
- Israel (7):
  - Research Site, Holon
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Tiberias
  - Research Site, Tzrifin
- Italy (8):
  - Research Site, Genova, GE
  - Research Site, Rozzano, MI
  - Research Site, Roma, Roma
  - Research Site, Ancona
  - Research Site, Genova
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rozzano
- Research Site, Riga, Latvia
- Malta (2):
  - Research Site, Floriana
  - Research Site, Valletta
- Philippines (4):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Molo
  - Research Site, Quezon City
- Poland (8):
  - Research Site, Bytom
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Rybnik
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Barnaul
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Tomsk
  - Research Site, Tyumen
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nitra
  - Research Site, Prešov
- South Africa (5):
  - Research Site, Lyttelton Manor, South Africa
  - Research Site, Cape Town
  - Research Site, Polokwane
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- Spain (19):
  - Research Site, Córdoba, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Barcelona, Catalonia
  - Research Site, Granollers, Catalonia
  - Research Site, Hospitalet de Llobregat(barcel, Catalonia
  - Research Site, Terrassa(barcelona), Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Valencia, Valencia
  - Research Site, A Coruña
  - Research Site, Córdoba
  - Research Site, Granollers
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Madrid
  - Research Site, Manresa
  - Research Site, Oviedo
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (3):
  - Research Site, Taoyuan District, Taiwan
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (6):
  - Research Site, Nakhonratchasima, Naimuang
  - Research Site, Chiang Mai, Thailand
  - Research Site, Songkhla, Thailand
  - Research Site, Chiang Mai
  - Research Site, Rachathewi
  - Research Site, Songkhla
- Turkey (Türkiye) (3):
  - Research Site, Istanbul, Goztepe
  - Research Site, Ankara
  - Research Site, Izmir
- Ukraine (17):
  - Research Site, Cherkassy
  - Research Site, Chernihiv
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Luhansk
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Simferopol
  - Research Site, Sumy
  - Research Site, Ternopil
  - Research Site, Uzhhorod
- United Kingdom (16):
  - Research Site, Southampton, Hampshire
  - Research Site, Maidstone, Kent
  - Research Site, Northwood, Middlesex
  - Research Site, Sutton, Surrey
  - Research Site, Bebington
  - Research Site, Bournemouth
  - Research Site, Bradford
  - Research Site, Guildford
  - Research Site, Ipswich
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Newcastle upon Tyne
  - Research Site, Northwood
  - Research Site, Poole
  - Research Site, Stockport
  - Research Site, Sutton
- Vietnam (4):
  - Research Site, Hanoi, Vietnam
  - Research Site, Ho Chi Minh City, Vietnam
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Abdel-Rahman O. Effect of Body Mass Index on 5-FU-Based Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer; A Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Dec;18(4):e385-e393. doi: 10.1016/j.clcc.2019.07.005. Epub 2019 Jul 15. PMID 31378656
- [Derived] Abdel-Rahman O. Impact of Sex on Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer: Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Jun;18(2):110-115.e2. doi: 10.1016/j.clcc.2018.12.006. Epub 2018 Dec 28. PMID 30679026
- [Derived] Robertson JD, Botwood NA, Rothenberg ML, Schmoll HJ. Phase III trial of FOLFOX plus bevacizumab or cediranib (AZD2171) as first-line treatment of patients with metastatic colorectal cancer: HORIZON III. Clin Colorectal Cancer. 2009 Jan;8(1):59-60. doi: 10.3816/CCC.2009.n.010. PMID 19203899
- See also: CSR-D8480C00013.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=417&filename=CSR-D8480C00013.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled = 1814 though not all patient randomised. Randomised= Intent to treat (ITT): Cediranib 20mg 709, Cediranib 30mg 192 Bevacizumab 713; Safety: Cediranib 20mg 705, Cediranib 30mg 191 Bevacizumab 704
Pre-assignment Details: Cediranib 30mg discontinued following Phase II, Cediranib 20mg chosen dose for comparing with Bevacizumab.
  200 patients dropped prior to treatment. Study was set up as a phase II/III study. Participants were enrolled into both phases if they participated in both Phase II/III, but are only counted once in the Enrollment Number and in the Results.
Groups:
- Cediranib 20 mg: Cediranib 20 mg/day + FOLFOX
  The FOLFOX regimen in this study was a modified FOLFOX6 regimen, repeated every 2 weeks:
  * Oxaliplatin 85 mg/m2 with leucovorin 400 mg/m2 (or equivalent folinic acid preparation) administered intravenously over 2 hours on Day 1
  * 5-FU 400 mg/m2 bolus immediately after completion of the oxaliplatin infusion on Day 1, followed immediately by 5-FU 2400 mg/m2 administered by a continuous iv infusion over 46 hours.
- Bevacizumab 5 mg/kg: Bevacizumab 5 mg/kg on Day 1 and every 2 weeks + FOLFOX
  The FOLFOX regimen in this study was a modified FOLFOX6 regimen, repeated every 2 weeks:
  * Oxaliplatin 85 mg/m2 with leucovorin 400 mg/m2 (or equivalent folinic acid preparation) administered intravenously over 2 hours on Day 1
  * 5-FU 400 mg/m2 bolus immediately after completion of the oxaliplatin infusion on Day 1, followed immediately by 5-FU 2400 mg/m2 administered by a continuous iv infusion over 46 hours.
- Cediranib 30 mg: Cediranib 30 mg/day + FOLFOX
  The FOLFOX regimen in this study was a modified FOLFOX6 regimen, repeated every 2 weeks:
  * Oxaliplatin 85 mg/m2 with leucovorin 400 mg/m2 (or equivalent folinic acid preparation) administered intravenously over 2 hours on Day 1
  * 5-FU 400 mg/m2 bolus immediately after completion of the oxaliplatin infusion on Day 1, followed immediately by 5-FU 2400 mg/m2 administered by a continuous iv infusion over 46 hours.
Period: Overall Study
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Started | 709 | 713 | 192
Completed | 397 | 394 | 60
Not Completed | 312 | 319 | 132
Not completed — Death | 239 | 247 | 105
Not completed — Withdrawal by Subject | 52 | 48 | 22
Not completed — Lost to Follow-up | 16 | 18 | 4
Not completed — Incorrect enrol/elig crit not fulfilled | 2 | 3 | 0
Not completed — Longer QTC as Visit 1 | 1 | 0 | 0
Not completed — Toxicity of treatment | 1 | 0 | 0
Not completed — Did not receive study treatment | 0 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Liver metastases, colon resec. planned | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg | Total
Number analyzed (Participants) | 709 | 713 | 192 | 1614
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 58.1 (11.37) | 59.0 (10.82) | 59.2 (10.59) | 58.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 297 | 299 | 73 | 669
    Male | 412 | 414 | 119 | 945

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression is defined as the number of months from randomisation until progressive disease based on RECIST (progression of target lesions, clear progression of existing non-target lesions or the appearance of one or more new lesions) or death in the absence of progression.
Time Frame: Baseline then at Weeks 8, 16, 24 and then every 12 weeks until progression
Population: Two cediranib doses (20 mg and 30 mg) were initially included in this study; however, it was intended that one dose would be selected for continuation. The decision was taken to continue with cediranib 20 mg. No statistical analyses were performed on the 30mg group.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Number analyzed (Participants) | 709 | 713 | 0
Months | 9.9 [6.3 to 13.5] | 10.3 [6.5 to 14.1] |

2. Secondary Outcome: Overall Survival
Description: Number of months from randomisation to the date of death from any cause
Time Frame: Randomisation until data cut-off
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Number analyzed (Participants) | 709 | 713 | 0
Months | 22.8 [13.3 to 32.3] | 21.3 [12.2 to 32.8] |

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate is Complete Response (CR) + Partial Response (PR) as defined below:
  CR = Disappearance of all target lesions. PR = At least a 30% decrease in the sum of longest diameters (LDs) of target lesions, taking as reference the baseline sum of LDs.
Time Frame: Up until data cut-off
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Number analyzed (Participants) | 709 | 713 | 0
Participants | 328 | 337 |

4. Secondary Outcome: Duration of Response
Description: Duration of Response is calculated as the time from the first recording of CR/PR until the patient progresses, regardless of whether the patient was still taking study medication. Only confirmed responses are included in the calculation. For patients who had not progressed, the end date used in the calculation of duration of response is the data cut-off date of 15th November 2009.
Time Frame: Up until data cut-off date of 15/11/2007
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Number analyzed (Participants) | 328 | 337 | 0
Months | 8.6 [6.1 to 12.1] | 9.6 [6.5 to 13.6] |

5. Secondary Outcome: Percentage Change in Tumour Size
Description: Percentage change in tumour size from baseline to first RECIST assessment (Week 8) ((Week 8 - baseline)/baseline)*100
Time Frame: Baseline to Week 8
Population: No statistical analyses were performed on the 30mg group. Patients had to have both a baseline and post-baseline (week 8) value to be included in the analysis. If patients did not have a week 8 assessment they were not included.
Measure: Mean (Standard Deviation); unit: Percentage change in tumour size
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Number analyzed (Participants) | 634 | 649 | 0
Percentage change in tumour size | -23.2 (21.8) | -22.1 (19.55) |

6. Secondary Outcome: Time to Worsening of Health Related Quality of Life (QOL) Based on the FACT Colorectal Symptom Index (FCSI)
Description: Time to worsening of symptoms, as measured by the FACT colorectal symptom index (FCSI), will be defined as the time when a sustained clinically important deterioration in the total score from the FCSI has been recorded.
Time Frame: Baseline through to data cut-off
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Cediranib 20 mg | Bevacizumab 5 mg/kg | Cediranib 30 mg
Number analyzed (Participants) | 709 | 713 | 0
Days | 170 [56 to 328] | 245 [112 to 348] |

ADVERSE EVENTS:
Groups:
- 1Bevacizumab 5mg/kg: Bevacizumab 5 mg/kg on Day 1 and every 2 weeks
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | 1Bevacizumab 5mg/kg
Serious Adverse Events (participants affected / at risk) | 275/705 | 90/191 | 231/704
Other Adverse Events (participants affected / at risk) | 684/705 | 187/191 | 672/704
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 20 mg (N=705) | Cediranib 30 mg (N=191) | 1Bevacizumab 5mg/kg (N=704)
Febrile Neutropenia (Blood and lymphatic system disorders) | 11 | 1 | 13
Neutropenia (Blood and lymphatic system disorders) | 8 | 5 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 0 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 3
Cardiac Failure (Cardiac disorders) | 3 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 3 | 1 | 2
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 2
Myocardial Infarction (Cardiac disorders) | 2 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Arteriospasm Coronary (Cardiac disorders) | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Atrial Thrombosis (Cardiac disorders) | 1 | 0 | 1
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1
Intracardiac Thrombus (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1 | 0
Pericarditis Constrictive (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Dihydropyrimidine Dehydrogenase Deficiency (Congenital, familial and genetic disorders) | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Diplopia (Eye disorders) | 1 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 30 | 11 | 13
Intestinal Obstruction (Gastrointestinal disorders) | 9 | 2 | 12
Vomiting (Gastrointestinal disorders) | 11 | 3 | 12
Abdominal Pain (Gastrointestinal disorders) | 9 | 2 | 10
Nausea (Gastrointestinal disorders) | 10 | 1 | 4
Ileus (Gastrointestinal disorders) | 7 | 2 | 6
Small Intestinal Obstruction (Gastrointestinal disorders) | 7 | 0 | 7
Stomatitis (Gastrointestinal disorders) | 7 | 2 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1 | 6
Rectal Haemorrhage (Gastrointestinal disorders) | 5 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 4
Constipation (Gastrointestinal disorders) | 3 | 1 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 3
Subileus (Gastrointestinal disorders) | 3 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colonic Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Periproctitis (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Reflux Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Varices Oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 21 | 9 | 11
Fatigue (General disorders) | 6 | 7 | 0
Asthenia (General disorders) | 3 | 2 | 1
Malaise (General disorders) | 3 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 3 | 2 | 1
Catheter Related Complication (General disorders) | 2 | 0 | 0
Catheter Thrombosis (General disorders) | 2 | 0 | 1
Chills (General disorders) | 2 | 0 | 0
Multi-Organ Failure (General disorders) | 2 | 0 | 0
Death (General disorders) | 1 | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 1 | 0
Infusion Site Extravasation (General disorders) | 1 | 0 | 0
Infusion Site Inflammation (General disorders) | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Sudden Death (General disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 2 | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Pain (Hepatobiliary disorders) | 0 | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 2 | 1 | 5
Hypersensitivity (Immune system disorders) | 0 | 0 | 2
Food Allergy (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 2 | 5
Catheter Related Infection (Infections and infestations) | 6 | 1 | 6
Sepsis (Infections and infestations) | 6 | 1 | 6
Urinary Tract Infection (Infections and infestations) | 6 | 1 | 3
Central Line Infection (Infections and infestations) | 4 | 0 | 4
Infection (Infections and infestations) | 4 | 0 | 1
Catheter Sepsis (Infections and infestations) | 1 | 0 | 3
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 3
Abscess (Infections and infestations) | 0 | 0 | 2
Anal Abscess (Infections and infestations) | 2 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Herpes Zoster (Infections and infestations) | 0 | 0 | 2
Septic Shock (Infections and infestations) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 2
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 2
Abdominal Abscess (Infections and infestations) | 0 | 1 | 0
Abdominal Infection (Infections and infestations) | 0 | 1 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0
Breast Abscess (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Catheter Site Cellulitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Clostridial Infection (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Enterococcal Infection (Infections and infestations) | 1 | 0 | 0
Gas Gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Gingival Infection (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Herpes Virus Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Infusion Site Infection (Infections and infestations) | 0 | 0 | 1
Liver Abscess (Infections and infestations) | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0
Mucormycosis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 0 | 1
Pelvic Abscess (Infections and infestations) | 1 | 0 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Retroperitoneal Abscess (Infections and infestations) | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Viral Diarrhoea (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 3 | 0 | 0
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac Valve Replacement Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Drug Toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 0
Blood Pressure Increased (Investigations) | 2 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0
Body Temperature Increased (Investigations) | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 1
Electrocardiogram Qt Prolonged (Investigations) | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 0
Glomerular Filtration Rate Decreased (Investigations) | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 1
Transaminases Increased (Investigations) | 0 | 0 | 1
Viral Test Positive (Investigations) | 1 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 5 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid Intake Reduced (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 3 | 2 | 1
Syncope (Nervous system disorders) | 3 | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 3 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Facial Palsy (Nervous system disorders) | 1 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0 | 1
Nerve Root Lesion (Nervous system disorders) | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 1 | 0
Partial Seizures (Nervous system disorders) | 0 | 0 | 1
Peroneal Nerve Palsy (Nervous system disorders) | 0 | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Toxic Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Vascular Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Dissociative Disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2
Renal Failure (Renal and urinary disorders) | 2 | 1 | 1
Bladder Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Renal Pain (Renal and urinary disorders) | 1 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 2
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 9 | 2 | 9
Hypertension (Vascular disorders) | 9 | 4 | 2
Jugular Vein Thrombosis (Vascular disorders) | 3 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 2 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 2
Arterial Thrombosis Limb (Vascular disorders) | 0 | 0 | 1
Circulatory Collapse (Vascular disorders) | 1 | 0 | 0
Embolism Venous (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 1
Shock Haemorrhagic (Vascular disorders) | 1 | 0 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Vasospasm (Vascular disorders) | 1 | 0 | 0
Vena Cava Thrombosis (Vascular disorders) | 1 | 1 | 1
Venous Thrombosis (Vascular disorders) | 1 | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 20 mg (N=705) | Cediranib 30 mg (N=191) | 1Bevacizumab 5mg/kg (N=704)
Neutropenia (Blood and lymphatic system disorders) | 302 | 85 | 228
Thrombocytopenia (Blood and lymphatic system disorders) | 186 | 55 | 85
Anaemia (Blood and lymphatic system disorders) | 50 | 16 | 79
Leukopenia (Blood and lymphatic system disorders) | 56 | 20 | 52
Hypothyroidism (Endocrine disorders) | 35 | 24 | 8
Diarrhoea (Gastrointestinal disorders) | 486 | 147 | 354
Nausea (Gastrointestinal disorders) | 355 | 100 | 349
Stomatitis (Gastrointestinal disorders) | 252 | 77 | 187
Vomiting (Gastrointestinal disorders) | 221 | 64 | 192
Constipation (Gastrointestinal disorders) | 145 | 34 | 187
Abdominal Pain (Gastrointestinal disorders) | 161 | 49 | 124
Abdominal Pain Upper (Gastrointestinal disorders) | 82 | 21 | 59
Dyspepsia (Gastrointestinal disorders) | 45 | 11 | 56
Dry Mouth (Gastrointestinal disorders) | 33 | 10 | 30
Dysphagia (Gastrointestinal disorders) | 22 | 11 | 10
Fatigue (General disorders) | 314 | 89 | 299
Pyrexia (General disorders) | 92 | 26 | 123
Asthenia (General disorders) | 96 | 31 | 73
Oedema Peripheral (General disorders) | 28 | 14 | 39
Drug Hypersensitivity (Immune system disorders) | 41 | 10 | 50
Nasopharyngitis (Infections and infestations) | 42 | 21 | 50
Urinary Tract Infection (Infections and infestations) | 42 | 15 | 43
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 4 | 36
Weight Decreased (Investigations) | 80 | 32 | 56
Alanine Aminotransferase Increased (Investigations) | 18 | 11 | 13
Decreased Appetite (Metabolism and nutrition disorders) | 177 | 71 | 160
Hypokalaemia (Metabolism and nutrition disorders) | 59 | 16 | 38
Back Pain (Musculoskeletal and connective tissue disorders) | 54 | 20 | 63
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 46 | 16 | 38
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 15 | 40
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 40 | 7 | 35
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 11 | 22
Neuropathy Peripheral (Nervous system disorders) | 218 | 49 | 212
Paraesthesia (Nervous system disorders) | 157 | 46 | 158
Peripheral Sensory Neuropathy (Nervous system disorders) | 135 | 37 | 144
Headache (Nervous system disorders) | 117 | 46 | 90
Dysgeusia (Nervous system disorders) | 82 | 24 | 84
Dizziness (Nervous system disorders) | 51 | 16 | 33
Lethargy (Nervous system disorders) | 40 | 12 | 30
Insomnia (Psychiatric disorders) | 49 | 16 | 55
Depression (Psychiatric disorders) | 23 | 11 | 23
Proteinuria (Renal and urinary disorders) | 48 | 23 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 169 | 45 | 172
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 124 | 47 | 81
Cough (Respiratory, thoracic and mediastinal disorders) | 71 | 22 | 68
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 60 | 27 | 43
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 44 | 13 | 37
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 104 | 31 | 68
Alopecia (Skin and subcutaneous tissue disorders) | 65 | 18 | 64
Rash (Skin and subcutaneous tissue disorders) | 51 | 14 | 38
Hypertension (Vascular disorders) | 292 | 92 | 183
Phlebitis (Vascular disorders) | 22 | 10 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.